CLINICAL TRIAL: NCT00696644
Title: An Italian Observational Study to Evaluate Fracture Outcomes, Compliance to Treatment, Back Pain, Health-related Quality of Life in Patients With Severe Osteoporosis Treated According to Common Clinical Practice
Brief Title: A Study for Teriparatide in Severe Osteoporosis
Acronym: ISSO
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 12456; B3D-IT-B014 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with severe osteoporosis: Postmenopausal women and men aged > 21 years old affected by severe osteoporosis
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — 20 mcg daily subcutaneous for 18 months.

SUMMARY:
This observational study will evaluate the incidence of new vertebral and non vertebral fragility fractures in patients with severe osteoporosis treated with anabolic drugs. This study will also evaluate BMD, compliance to treatment, back pain and the health-related quality of life.

DETAILED DESCRIPTION:
The participants should be treated with anabolic therapy for osteoporosis (Teriparatide or PTH 1-84) for 18 months and should be followed up for subsequent 6 months. The treatment is expected to improve bone mineral density, back pain and reduce the risk of new fractures due to osteoporosis. The outcomes will be evaluated by bone densitometry at the lumbar spine and femoral neck, by standard radiographs, by measurements of bone formation marker (P1NP) and by questionnaires on back pain and quality of life. Postmenopausal women and men over 21 years old may be included if they have:

1. at least 3 severe vertebral fractures
2. 2 severe vertebral fractures and 1 hip fracture
3. an incidental vertebral fracture or an hip fracture during treatment with antiresorptives prescribed for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women and men older than 21 years affected by severe osteoporosis with an incidental vertebral or hip fracture during treatment with an antiresorptive, or having 3 or more severe vertebral fractures or having 2 severe vertebral fractures and an historical hip fracture.

Exclusion Criteria:

* Any contraindication for the use of antiosteoporotic drug
* Premenopausal women or men younger than 21 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 794 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of any osteoporotic fractures in the first 24 months from the initiation of anabolic medication. | From 0 to 24 months

SECONDARY OUTCOMES:
Treatment compliance | From 0 to 24 months
Reason of discontinuation | From 0 to 24 months
BMD changes (lumbar and femoral BMD) | From 0 to 24 months
Changes in bone turnover marker measured by P1NP | From 0 to 24 months
Quality of Life (measured by EQ-5D of EuroQol Group) | From 0 to 24 months
Back Pain measured by visual analogue scale and back pain questionnaire | From 0 to 24 months
Assessment of motor performance and chair rising test | From 0 to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this study, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valeggio sul Mincio, Verona, Italy

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com